CLINICAL TRIAL: NCT04133675
Title: A Single-Blind, Randomized Study of the BTL EmsellaTM Chair Versus Sham for the Treatment of Stress Urinary Incontinence
Brief Title: BTL Emsella Chair Versus Sham for the Treatment of Stress Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-242
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence
Keywords: urinary incontinence; urine leakage
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive active Emsella chair treatments or sham treatments. Study will be performed in a single-blind manner.(Participant and biostatistician)
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be performed using a table of random numbers. A unblinded RNC will be responsible for maintaining the enrollment and randomization log. Randomization envelopes will be provided by the study's biostatistician and will be securely stored in a locked cabinet. The study coordinator(s) will solely be responsible for opening the randomization envelopes and delivering the study treatments, according to group assignment. Ultimately, they will be responsible for maintaining the confidentiality and security of the randomization envelopes. After randomization, the study coordinator(s) will complete the Subject Enrollment and Randomization Log. The log may be stored in a locked cabinet with the randomization envelopes. At study completion the log will be stored in the regulatory binder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Emsella Chair Active Treatment (Active Comparator): Active treatment subjects will be asked to sit on the center of the Emsella chair. The height of the chair will be adjusted until the participant's feet are on the floor. The Emsella chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will then be decreased slightly and stay unchanged for the remainder of the treatment time. The treatment threshold should be increased with every treatment until the subject reaches 100%.
  Interventions: Device: BTL Emsella
- Emsella Sham Treatment (Sham Comparator): Sham subjects will be positioned on the device in the same manner as the active treatment group. The sham treatment will be provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below therapeutic level (<10% power).
  Interventions: Device: Sham BTL Emsella

INTERVENTIONS:
Device: BTL Emsella — The Emsella Chair is a novel high-intensity focused electromagnetic (HIFEM) technology for the treatment of SUI, in addition to other pelvic floor related disorders. HIFEM technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercises over 28 minutes. The treatment paradigm consists of 3 different phases. The phases consist of an intense stimulation of the pelvic floor muscles (PFM), which consists of stimlulation and relaxation. The repetition of the phases and focused electromagnetic energy delivery leads to pelvic floor stimulation, adaptation, and remodelation.
  Arms: Emsella Chair Active Treatment
Device: Sham BTL Emsella — Sham subjects will be positioned on the device in the same manner as the active treatment group. The sham treatment will be provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below therapeutic level (<10% power).
  Arms: Emsella Sham Treatment

SUMMARY:
Stress urinary incontinence (SUI) is a condition that affects both men and women. SUI is the involuntary leakage of urine caused by an increase in intra-abdominal pressure from activities such as exercise, coughing, laughing, or sneezing. It can significantly affect quality of life as patients avoid activities or behaviors that cause leakage. This clinical trial will compare the efficacy of the Emsella chair to sham and determine if electromagnetic technology is effective in the treatment of SUI.

DETAILED DESCRIPTION:
This is a prospective, sham-controlled, observational study of subjects undergoing electromagnetic perineal stimulation for the treatment of SUI. Eligible subjects will be randomized to receive active treatment or sham in a 1:1 ratio. Eight treatments (2 treatments each week) for 4 weeks will be completed with the Emsella chair to the pelvic floor muscles.

Electromagnetic stimulation of the pelvic floor is a FDA approved therapy whereby a coil generates pulsed electromagnetic fields that penetrate deep into the pelvic floor muscles inducing stimulation and providing rehabilitation of weak pelvic muscles.The Emsella Chair is a novel high-intensity focused electromagnetic (HIFEM) technology for the treatment of SUI, in addition to other pelvic floor related disorders. HIFEM technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercises over 28 minutes.This technology is typically not covered by insurance, is minimally invasive, and safe, but has limited data available.

Currently, there is no data available from sham controlled studies evaluating efficacy of this technology. The purpose of this study is to compare the Emsella Chair to sham and to determine whether electromagnetic technology is effective in the treatment of SUI.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written, dated, informed consent prior to screening, and be likely to comply with study protocol, including independently complete study questionnaires and communicate with study personnel about AEs and other clinically important information.
2. Females and males, 18 to 80 years of age, inclusive, at screening
3. Positive Cough or Bladder Stress Test at screening
4. Subject agrees not to start any new treatment (medication or otherwise) during the treatment and follow-up periods.

6. Subject agrees to maintain a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, beta-3 adrenergic agonist, or α-adrenergic blockers, throughout the treatment and follow-up periods.

For Females Only:

* Subject agrees to discontinue use of bladder support devices, including but not limited to vaginal pessary, during the screening, treatment, and follow-up periods.
* If of child-bearing age and female, agree to practice approved birth-control methods (oral contraceptives, condom barrier, injection, diaphragm or cervical cap, vaginal contraceptive ring, IUD, implantable contraceptive, surgical sterilization (bilateral tubal ligation), vasectomized partner(s))

For Males Only:

- Subject must be ≥ 4 months post radical prostatectomy

Exclusion Criteria:

1. Pelvic floor physical therapy, including muscle training and/or electrostimulation, in a clinical setting within 30 days prior to screening
2. Subject is morbidly obese (defined as body mass index 40 or greater)
3. Pulmonary insufficiency, defined as difficulty breathing and fatigue, especially during exercise; chest pain, such as squeezing, pressure or tightness; the sensation of rapid or irregular heartbeat (palpitations); swelling of the legs or feet; dizziness or fainting; and/or bluish discoloration of the nails and/or lips (cyanosis)
4. Any condition that causes a lack of normal skin sensation to the pelvis, buttocks, and lower extremities
5. Implanted cardiac pacemaker or metal in the body, including, but not limited to drug pumps, neurostimulators, electronic implants, copper intrauterine devices (IUDs), and/or defibrillators
6. Subject has a piercing between the waist and knees and is not willing to remove it before each treatment
7. Active urethral diverticula
8. Known vesicoureteral reflux
9. Currently healing from surgical procedures where muscle contraction may disrupt the healing process
10. Treatment with urethral bulking agents within the 6 months prior to the Screening Visit
11. Subject is currently receiving treatment for a malignant tumor that would interfere with study participation.
12. Subject has used the BTL EMSELLA device previously
13. Subject has urinary incontinence of neurogenic etiology, such as multiple sclerosis, spina bifida, Parkinson's, spinal cord injury, diabetic neuropathy etc.
14. Clinically confirmed urinary tract infection, requiring treatment as determined by the investigator, at the Screening Visit
15. Currently participating in an investigational study that may impact study results or previously received an investigational drug or treatment within 30 days of the Screening Visit
16. Current or history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation

    For Females Only:
17. Pregnant, or planning to become pregnant, at screening or anytime throughout the study period
18. History of surgery with insertion of vaginal mesh for SUI
19. Vaginal prolapse beyond the introitus
20. Vaginal rejuvenation treatment, including laser treatments and radiofrequency therapy, within the 6 months prior to the Screening Visit

    * Note for the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence. | 4 weeks after completing all treatments
  The primary objective of this study is to compare the efficacy of Emsella Chair to sham by evaluating the the responder rate, where a patient is called a responder if there is ≥ 50% reduction from baseline in the number stress incontinence events.

SECONDARY OUTCOMES:
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence in relation to the change in total number of subject-reported stress urinary incontinence (SUI) episodes. | 8 weeks after completing all treatments
  Change in the total number of subject-reported stress incontinence (SUI) episodes over 3 days based on voiding diaries. Patients will be giving a 3-day void diary to complete.
The efficacy of the Emsella chair versus sham to treat SUI in relation to the change in subject-reported impression of SUI severity. | 8 weeks after completing all treatments
  Change in subject-reported impression of SUI severity as measured by the Patient Global Impression of Severity scale (PGI-S). The subject will check the box that describes how their condition is now. The available options are normal, mild, moderate, or severe.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence in relation to the change in subject-reported impression of SUI improvement as measured by the Patient Global Impression of Improvement scale (PGI-I). | 8 weeks after completing all treatments
  Change in subject-reported impression of SUI improvement as measured by the Patient Global Impression of Improvement scale (PGI-I). The subject will select one of the following options, (very much better, much better, a little better, no change, a little worse, much worse, very much worse) to describe their urinary tract symptoms now versus prior to study treatment.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence related to the change in subject-reported urogenital distress. | 8 weeks after completing all treatments
  Change in subject-reported urogenital distress as measured by the Urinary Distress Inventory questionnaire (UDI-6). The UDI-6 is a six point questionnaire, each question answered is scored as follows; 0 = no, 1 = not at all, 2 = somewhat, 3 = moderately, 4 = quite a bit. Add all scores and divide by 6, then multiply by 25 to calculate the raw score. Higher scores = higher disability.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence in relation to the change in subject-reported impact of SUI on daily life. | 8 weeks after completing all treatments
  Change in subject-reported impact of SUI on daily life as measured by the Incontinence Impact Questionnaire (IIQ-7) Short Form. The IIQ-7, assesses how their problem effects activities, relationships, and feelings. It is a 7 point questionnaire. Each answer is scored on the following scale 0 = not at all, 1 = slightly, 2 = moderately, 3 = greatly. The higher the score the more effected they are by their condition.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence in relation to the change in subject-reported impact of urinary incontinence on daily life measured by the Incontinence Quality of Life questionnaire (I-QOL). | 8 weeks after completing all treatments
  Change in subject-reported impact of urinary incontinence on daily life as measured by the Incontinence Quality of Life questionnaire (I-QOL). The I-QOL is a quality of life measure specific to persons with urinary incontinence. The survey consists of 22 incontinent-specific quality of life items all having the following five-point ordinal response; 1 = extremely, 2 = quite a bit, 3 = moderately, 4 = a little, 5 = not at all. The summed total score is transformed to a 0-100 scale ranging from 0 (poor quality of life) to 100 (maximum quality of life).
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence and the change in fecal incontinence as measured by the Cleveland clinic incontinence score (Wexner). | 8 weeks after completing all treatments
  Change in subject-reported fecal incontinence as measured by the Cleveland clinic incontinence score (Wexner). The type of incontinence of stool (solid, liquid, gas, wears pad, lifestyle altered) are reported by the subject. Each question is measured as 0 = never, 1 = rarely, 2 = sometimes, 4 = usually, 5 = always. The higher the score the more severe the condition.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence and the change in subject-reported sexual function as measured by Female Sexual Function Index questionnaire for female subjects. | 8 weeks after completing all treatments
  The change in subject-reported sexual function as measured by the Female Sexual Function Index questionnaire (FSFI) for female subjects. The FSFI is a 19 question survey. A lower the score is equivalent a higher degree of sexual function. Scores range from 0 to 95.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence and the change in subject-reported sexual function as measured by the Brief Sexual Function Inventory questionnaire (BSFI) for male subjects. | 8 weeks after completing all treatments
  Change in subject-reported sexual function as measured by the Brief Sexual Function Inventory questionnaire (BSFI) for male subjects. The BSFI is a validated questionnaire for male sexual function. Scores range from 0 to 44. A lower score indicates a higher degree of dysfunction.
The efficacy of the Emsella chair versus sham to treat stress urinary incontinence and change in reported pain and discomfort. | 8 weeks after completing all treatments
  Change in subject-reported pain and discomfort as measured by the Visual Analog Scale (VAS). The VAS is a validated questionnaire that assesses pain on a scale from 0 = no pain to 10 = Worst possible pain.
Durability to determine whether subjects in the Emsella Chair group continue to have a higher responder rate than the Sham group | 8 weeks after primary efficacy endpoint
  The secondary object for durability for this study are to determine whether subjects in the Emsella Chair group continue to have a higher responder rate than the Sham group
Safety objective to determine the safety and tolerability of Emsella Chair compared to sham | 4 weeks after primary efficacy endpoint
  Safety and tolerability of the Emsella chair compared to Sham will be assessed in relation the incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galloway NT, El-Galley RE, Sand PK, Appell RA, Russell HW, Carlan SJ. Extracorporeal magnetic innervation therapy for stress urinary incontinence. Urology. 1999 Jun;53(6):1108-11. doi: 10.1016/s0090-4295(99)00037-0. PMID 10367836
- [Background] HIFEM technology in treatment of urinary incontinence mechanism of action. https://www.avantemedicalcenter.com/images/documents/Emsella_study.pdf. Published November 2017. Accessed June 20, 2019.